CLINICAL TRIAL: NCT01290991
Title: A Pilot Study to Augment™ Bone Graft Plus Evaluate the Safety of Allograft for Treatment of Osteochondral Defects (OCD) of the Knee
Brief Title: A Study to Evaluate the Safety of Augment™ Bone Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, William Stanish, Medical Doctor, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stanish-2010-01
Record Dates: First submitted 2011-02-02; First posted 2011-02-07 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Defect of Articular Cartilage
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone Graft (Other): Single Arm.. Augment Bone Graft for Osteochondral Defects
  Interventions: Device: Augment Bone Graft

INTERVENTIONS:
Device: Augment Bone Graft — Augment Bone Graft physically fills bone defects by providing a biocompatible scaffold for new bone formation.The material is comprised of a matrix of beta tricalcium phosphate and a highly purified recombinant human platelet-derived growth factor.
  Other Names: Bone Graft

SUMMARY:
Is Augment Bone Graft plus Allograft safe to use for the treatment of osteochondral defects of the knee?

DETAILED DESCRIPTION:
Subjects will be 18 to 40 years with an osteochondral defects of the knee.They will be candidates for allograft and Augment Bone Graft will be added to the procedure. The safety of Augment Bone Graft plus allograft for osteochondral defects of the knee will be evaluated by type, frequency, severity and relatedness of adverse events to the device for a minimum of 24 weeks.Magnetic Resonance Imaging will be performed at 1,12 and 42 weeks to evaluate device integrity and surgical treatment of osteochondral defects. Computed tomography will be done at week 1 and week 24 to determine the healing status of the osteochondral defect.

ELIGIBILITY:
Inclusion Criteria:

* Prior Magnetic Resonance Imaging (MRI) evaluation or MRI on Screening.
* Subjects with Grade III osteochondral defect (OCD) of femoral condyle.
* Subjects with OCD > 1 cm.squared.
* Independent and ambulatory pts.
* Subjects from 18 to 40 years of age.
* Subject with a stable knee joint and similar stability on the opposite knee.
* Subject has knee x-ray with < 15 degrees of valgus and < 5 degrees varus.
* No deformity from previous fractures of tibia or fibula.
* BMI < 35.
* Subject has an American Association of Anaesthetists physical status classification of 1 or 2.
* Subject must present with pain > 3.0 cm according to the Visual Analogue Score.
* Subject has exhausted non operative treatment.

Exclusion:

* Allergy to yeast derived products.
* Index knee has had cartilage repair in the last six months.
* Subjects with osteoarthritis,inflammatory arthritis, rheumatoid arthritis and avascular necrosis of index knee.
* Subject has contralateral knee complications which would interfere with rehabilitation
* Subject has implanted metallic devices that would prevent Magnetic Resonance Imaging (MRI).
* Subject has claustrophobia that would prevent MRI.
* Subject has had a malignancy or is being treated for a malignancy.
* Subject is physically or mentally compromised that would interfere with compliance.
* Subject is a prisoner or transient.
* Subject has a recent history (12 months) of alcohol abuse.
* Subject is pregnant, able to become pregnant but not practising birth control.
* Subject has an infection in the operative area.
* Subject has scheduled surgery on the contralateral knee over the course of the study.
* Subject requires another procedure in the index knee.
* Subject has had steroid therapy in the past six months.
* Subject is taking prescription pain medication for another indication other than the index knee.
* Subject is using nicotine in any form.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of Augment Bone Graft plus Allograft for treatment of osteochondral defects of the knee. | 12 months
  Collection of related adverse events

SECONDARY OUTCOMES:
To utilize Magnetic Resonance Imaging to evaluate device integrity and surgical treatment of osteochondral defects of the knee. | 12 months
  Assess healing and bone formation from radiological reports

CONTACTS AND LOCATIONS:
Overall Officials: William D Stanish, MD, Principal Investigator — Capital Dictrict Health Authority
Locations (1):
- Queen Elizabeth ll Health Sciences Centre, Halifax, Nova Scotia, Canada